CLINICAL TRIAL: NCT00121303
Title: Randomised Induction and Post Induction Therapy in Older Patients (≥61 Years of Age) With Acute Myeloid Leukemia (AML) and Refractory Anemia With Excess Blasts (RAEB, RAEB-t)
Brief Title: Cytarabine and Daunorubicin With or Without Gemtuzumab Ozogamicin in Treating Older Patients With Acute Myeloid Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000433422; SAKK-AML-43; EU-20514; HOVON-AML-43
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; secondary acute myeloid leukemia; untreated adult acute myeloid leukemia; de novo myelodysplastic syndromes; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Anemia, Refractory, with Excess of Blasts; Congenital Abnormalities | interventions — Cytarabine; Daunorubicin; Gemtuzumab

ARMS (4):
- Arm A low dose Dauno (Active Comparator): Induction 45 mg Dauno
  Interventions: Drug: cytarabine; Drug: daunorubicin hydrochloride
- ARM B high dose Dauno (Experimental): Induction 90 mg Dauno
  Interventions: Drug: cytarabine; Drug: daunorubicin hydrochloride
- Arm 1 no further treatment (No Intervention)
- Arm 2 Mylotarg (Experimental): Post induction treatment with Mylotarg
  Interventions: Drug: gemtuzumab ozogamicin

INTERVENTIONS:
Drug: cytarabine
  Arms: ARM B high dose Dauno; Arm A low dose Dauno
Drug: daunorubicin hydrochloride
  Arms: ARM B high dose Dauno; Arm A low dose Dauno
Drug: gemtuzumab ozogamicin
  Arms: Arm 2 Mylotarg

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine and daunorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as gemtuzumab ozogamicin, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether cytarabine and daunorubicin followed by gemtuzumab ozogamicin is more effective than cytarabine and daunorubicin in treating acute myeloid leukemia or myelodysplastic syndromes.

PURPOSE: This randomized phase III trial is studying cytarabine and two different doses of daunorubicin to see how well they work compared to cytarabine and daunorubicin followed by gemtuzumab ozogamicin in treating older patients with acute myeloid leukemia or myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the event-free and disease-free survival of older patients with acute myeloid leukemia, refractory anemia with excess blasts (RAEB), or RAEB in transformation treated with induction therapy comprising cytarabine in combination with two different doses of daunorubicin followed by cytarabine alone with or without post-induction therapy comprising gemtuzumab ozogamicin.

Secondary

* Compare the complete remission rate in patients treated with these regimens.
* Compare the overall survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Determine the probability of relapse and death during first complete remission in patients treated with post-induction gemtuzumab ozogamicin.
* Correlate prognostic factors (e.g., CD33 positivity, multidrug resistance phenotype, or cytogenetics) with probability of complete remission and overall, event-free, and disease-free survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and diagnosis (acute myeloid leukemia [AML] vs myelodysplastic syndromes [MDS]) for induction therapy. Patients are stratified according to participating center, diagnosis (AML vs MDS), induction treatment arm (I vs II), and response to induction therapy (complete remission [CR] vs no CR) for post-induction therapy.

* Induction therapy (course 1): Patients are randomized to 1 of 2 induction treatment arms.

  * Arm I: Patients receive cytarabine IV continuously on days 1-7 and daunorubicin IV over 3 hours on days 1-3.
  * Arm II: Patients receive cytarabine as in arm I and daunorubicin as in arm I but at a higher dose.

Approximately 28-35 days after the start of course 1 (or sooner if the bone marrow shows evidence of resistant disease), patients in both arms proceed to course 2 of induction therapy.

* Induction therapy (course 2): All patients receive cytarabine IV over 6 hours twice daily on days 1-6.

After completion of course 2, patients undergo assessment of remission status. Patients who do not achieve CR are removed from the study. Patients achieving CR proceed to post-induction therapy and undergo a second randomization.

* Post-induction therapy: Patients are randomized to 1 of 2 post-induction treatment arms.

  * Arm I: Patients receive no further chemotherapy.
  * Arm II: Patients receive gemtuzumab ozogamicin IV over 2 hours on days 1, 29, and 57 in the absence of disease relapse or unacceptable toxicity.

After completion of study treatment, patients are followed monthly for 1 year, every 3 months for 2 years, every 4-6 months for 2 years, and then periodically thereafter.

PROJECTED ACCRUAL: A total of 600 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML)

    * M0-M2 or M4-M7 FAB subtype

      * No AML with cytogenetic abnormality t(15;17) (M3)
    * Patients with secondary AML progressing from prior myelodysplasia* or biphenotypic leukemia are eligible
  * Refractory anemia with excess blasts (RAEB) or RAEB in transformation

    * International Prognostic Scoring System score ≥ 1.5 NOTE: *Any prior hematological disease of ≥ 4 months duration
* No chronic myelogenous leukemia in blastic crisis
* No prior polycythemia rubra vera
* No primary myelofibrosis

PATIENT CHARACTERISTICS:

Age

* 61 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* ALT and/or AST ≤ 2.5 times upper limit of normal (ULN)*
* Bilirubin ≤ 2 times ULN* NOTE: *Unless elevation is caused by organ infiltration by AML

Renal

* Creatinine ≤ 2 times ULN* NOTE: *Unless elevation is caused by organ infiltration by AML

Cardiovascular

* No myocardial infarction within the past 6 months
* LVEF > 50% by MUGA, echocardiogram, or other methods
* No unstable angina
* No unstable cardiac arrhythmia
* No severe and/or uncontrolled hypertension

Other

* No uncontrolled diabetes
* No severe and/or uncontrolled infection
* No other severe and/or uncontrolled medical condition

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 6 months since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior induction therapy for AML or myelodysplastic syndromes

Ages: 61 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Event-free survival after induction therapy
Disease-free survival after maintenance therapy

SECONDARY OUTCOMES:
Complete remission (CR) rate after induction therapy
Overall survival after induction therapy
Toxicity after induction therapy
Toxicity after maintenance therapy
Probability of relapse and death in first CR after maintenance therapy
Overall survival after maintenance therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kell, MRCPath, Study Chair — University Hospital of Wales
Locations (6):
- United Kingdom (6):
  - North Hampshire Hospital, Basingstoke, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Medway Maritime Hospital, Gillingham Kent, England
  - Maidstone Hospital, Maidstone, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - University Hospital of Wales, Cardiff, Wales